CLINICAL TRIAL: NCT04894942
Title: Evaluation of Clinical Features and Surgical Outcomes of the Too Long Anterior Process in Children: a Prospective Study
Brief Title: Evaluation of Clinical Features and Surgical Outcomes of the Too Long Anterior Process in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: Ballouhey _anterior process
Record Dates: First submitted 2021-05-09; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-03

CONDITIONS: Calcaneonavicular Coalition
MeSH Terms: conditions — Synostoses, tarsal, carpal, and digital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: American Orthopaedic Foot and Ankle Society Score (AOFASS) — calculation of the score AOFASS before and after the surgery

SUMMARY:
Calcaneonavicular coalition represents approximately 1% of the population between 8 and 12 years. They are manifested by repeated ankle sprains or by pain. - The diagnosis is radiological on an X-ray of the foot in oblique-3/4 incidence as well as magnetic resonance imaging. Treatment is second-line surgery after failure of orthopedic treatment. This surgery is either by direct approach or by arthroscopy, by performing a bone resection to recreate sufficient space in the joint in question. The patients in this study will only be operated on openly.

ELIGIBILITY:
Inclusion Criteria:

* Child <16 years
* Child with calcaneonavicular coalition
* Magnetic resonance imaging diagnosis
* Patient already treated orthopedically in the initial treatment of the coalition

Exclusion Criteria:

* Child >=16 years

Ages: 8 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Child <16 years with calcaneonavicular coalition with Magnetic resonance imaging diagnosis and already treated orthopedically in the initial treatment of the coalition
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of scores before surgery and after surgery at 1 month, for all the operated patients | 1 month
  Calculation of the American Orthopaedic Foot and Ankle Society Score. This is an instrument for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part.
  The maximal score is 100 points, indicating no symptoms or impairments.
Comparison of scores before surgery and after surgery at 3 months for all the operated patients | 3 months
  Calculation of the American Orthopaedic Foot and Ankle Society Score. This is an instrument for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part.
  The maximal score is 100 points, indicating no symptoms or impairments.
Comparison of scores before surgery and after surgery at 1 12 months for all the operated patients | 12 months
  Calculation of the American Orthopaedic Foot and Ankle Society Score. This is an instrument for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It combines a clinician-reported and a patient-reported part.
  The maximal score is 100 points, indicating no symptoms or impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric emergency department, Limoges, France